CLINICAL TRIAL: NCT03100708
Title: Evaluation of Molecular and Pathophysiological Mechanisms of Peritoneal Carcinomatosis and Monitoring of the Efficiency of PIPAC (Pressurized Intra-peritoneal Aerosol-Chemotherapy) as a Local Chemotherapeutical Treatment.
Brief Title: Register Study of Patients With Peritoneal Carcinomatosis Treated With PIPAC (Pressurized Intra-peritoneal Aerosol-Chemotherapy)
Acronym: PIPAC_01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. Boris Jansen-Winkeln, Dr. B. Jansen-Winkeln and Prof. Dr. I. Gockel, University of Leipzig
Other Study IDs: PIPAC_01
Record Dates: First submitted 2016-11-15; First posted 2017-04-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with peritoneal carcinomatosis: Patient with peritoneal carcinomatosis and the Indication for local therapy. The Clinics tumor-board advice is needed.
  Interventions: Procedure: PIPAC

INTERVENTIONS:
Procedure: PIPAC — * Cisplatin 7.5 mg/m2 body surface in 150 ml NaCl 0,9% + Doxorubicin 1.5 mg/m2 body surface in 50 ml NaCl 0,9% in patients with ovarian, gastric, pancreatic cancer and in primary peritoneal tumors.
  * Oxaliplatin 92 mg/m2 body surface in 150 ml dextrose solution in patients with colorectal cancer.
  The chemotherapeutics will be admitted to the abdomen by a nebulizer at a pressure of 200 psi and 12 mmHG with 0.5 mL/sec. Afterwards the chemotherapeutics can react for 30min before the abdominal gas will be drained to the clinics filtering system.
  Other Names: Pressurized Intra-peritoneal Aerosol-Chemotherapy

SUMMARY:
The study will follow up patients with peritoneal carcinomatosis from colorectal, ovarian, gastric, pancreatic cancers and primary peritoneal tumors and undergoing a diagnostic laparoscopy / laparotomy, a PIPAC as single dose or repeated every 6 weeks. The Overall Response Rate (ORR), the Overall Survival (OS) and the Quality of Life will be assessed before every PIPAC. Biopsies of the peritoneal carcinomatosis and blood (plasma and serum) are collected with every PIPAC intervention to follow up and to document the individual success or progress of the patients. The advice of the tumor board is mandatory to confirm the indication for local chemotherapy (PIPAC).

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical and pathological confirmed peritoneal carcinomatosis from gastric, colorectal, pancreatic, ovarian cancers or primary peritoneal tumors
* Age > 18 years
* signed informed consent

Exclusion Criteria:

* Patient can not understand meaning and purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffer from peritoneal carcinomatosis.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (years) | 5 years

SECONDARY OUTCOMES:
The Peritoneal Carcinomatosis Index (PCI) before and after repeated PIPAC treatments | 25 weeks
Overall Response Rate (CT RESIST criteria) | 5 years
  Complete response
Quality of lfe questionnaire (EORTC QLQ-C15-PAL) | 5 years
  Groenvold M et al. The development of the EORTC QLQ-C15-PAL: a shortened questionnaire for cancer patients in palliative care. European Journal of Cancer 2006; 42(1): 55-64

CONTACTS AND LOCATIONS:
Overall Officials: Ines Gockel, Prof. Dr., Principal Investigator — Universitätsklinikum Leipzig
Locations (1):
- Universitätsklinikum Leipzig - AöR, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jansen-Winkeln B, Eberth J, Moulla Y, Mehdorn M, Niebisch S, Schierle K, Blaker H, Lordick F, Gockel I, Thieme R. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) in patients with peritoneal surface malignancies (PSM): a prospective single-center registry study. J Cancer Res Clin Oncol. 2023 Mar;149(3):1331-1341. doi: 10.1007/s00432-022-04517-w. Epub 2022 Dec 13. PMID 36513815
- [Derived] Gockel I, Jansen-Winkeln B, Haase L, Niebisch S, Moulla Y, Lyros O, Lordick F, Schierle K, Wittekind C, Thieme R. Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) in patients with peritoneal metastasized colorectal, appendiceal and small bowel cancer. Tumori. 2020 Feb;106(1):70-78. doi: 10.1177/0300891619868013. Epub 2019 Aug 30. PMID 31469058
- [Derived] Gockel I, Jansen-Winkeln B, Haase L, Rhode P, Mehdorn M, Niebisch S, Moulla Y, Lyros O, Lordick F, Schierle K, Wittekind C, Thieme R. Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) in Gastric Cancer Patients with Peritoneal Metastasis (PM): Results of a Single-Center Experience and Register Study. J Gastric Cancer. 2018 Dec;18(4):379-391. doi: 10.5230/jgc.2018.18.e37. Epub 2018 Dec 14. PMID 30607301